CLINICAL TRIAL: NCT01978860
Title: A Prospective, First in Man Study to Evaluate the Safety and Performance of the NovaCross™ Micro-catheter in (CTO) Coronary Lesions
Brief Title: A Prospective, First in Man Study to Evaluate the Safety and Performance of the NovaCross™ Micro-catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chanan Schneider (Industry)
Collaborators: Clinical Research Consultants, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chanan Schneider, COO, Nitiloop Ltd.
Organization: Nitiloop Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-C200-02 Rev 01; HTA6696 (Other: Israeli Ministry of Health Department)
Record Dates: First submitted 2013-10-23; First posted 2013-11-08 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: CABG Coronary artery bypass grafting; CTO Chronic Total Occlusion; PCI Percutaneous coronary intervention; MACE Major adverse cardiovascular event(s); MI Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NovaCross, CTO (Experimental): assess the safety and technical feasibility, deployment and withdrawal characteristics of the NovaCross™ micro-catheter during an interventional coronary angioplasty procedure and evaluating the CTO penetration rate.
  Interventions: Device: NovaCross, CTO

INTERVENTIONS:
Device: NovaCross, CTO — evaluate the safety and performance of the NovaCross™ micro-catheter in respect to providing additional guidewire support that is expected to allow easier crossing of Chronic Total Occlusion (CTO) lesions in coronary arteries.

SUMMARY:
This is a prospective, non-randomized, first-in-man investigational study, to assess the safety and technical feasibility, deployment and withdrawal characteristics of the NovaCross™ micro-catheter during an interventional coronary angioplasty procedure and evaluating the CTO penetration rate.

Each study subject/patient will have a total of one (1) procedure performed for this study.

DETAILED DESCRIPTION:
To be filled later

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 25-80
2. Patient understands and has signed the study informed consent form.
3. Patient has an angiographic documented Chronic Total Occlusion (i.e. >3 months occlusion duration) showing distal TIMI flow 0.
4. Suitable candidate for non-emergent, coronary angioplasty
5. Documented coronary angiography preceding the PCI reveals at least one CTO lesion situated in a non-infarct related coronary artery or its side branches with the following characteristics:

   1. Thrombolysis in Myocardial Infarction (TIMI) 0 flow for at least 90 days;
   2. Satisfactory distal vessel visualization
   3. CTO should be amenable to percutaneous treatment and must be located in a coronary vessel with a reference diameter of at least 2 millimeters.
   4. CTO refractory to a minimum of 10 minutes of conventional guide wire attempt.
6. Body Mass Index (BMI) < 40
7. Left ventricle ejection fraction > 25%

For the purpose of this trial, a CTO is defined as a 100% luminal narrowing without antegrade flow or with antegrade or retrograde filling through collateral vessels.

-

Exclusion Criteria:

* 1. Patient unable to give informed consent. 2. Current participation in another study with any investigational drug or device.

  3. Patient is known or suspected not to tolerate the contrast agent. 4. Aorto-ostial CTO location (Ostial bifurcation origins may be considered), SVG CTO and in-stent CTOs.

  5. Intolerance to aspirin or Clopidogrel or Prasugrel or Ticagrelor medications 6. Appearance of a fresh thrombus or intraluminal filling defects. 7. Recent major cerebrovascular event (history of stroke or TIA within 1 month) 8. Cardiac intervention within 4 weeks of the procedure 9. Renal insufficiency (serum creatinine of > 2.3mg/dl) 10. Active gastrointestinal bleeding 11. Active infection or fever that may be due to infection 12. Life expectancy < 2 years due to other illnesses 13. Significant anemia (hemoglobin < 8.0 mg / dl) 14. Severe uncontrolled systemic hypertension (> 240 mmHg within 1 month of procedure )

  15. Severe electrolyte imbalance 16. Congestive heart failure [New York Heart Association (NYHA) Class III\IV] ,CSA Class IV.

  17. Unstable angina requiring emergent percutaneous trans-luminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) 18. Recent myocardial infarction (MI) (within the past two weeks) 19. Uncontrolled diabetes >2 serum glucose concentrations of >350 mg/dl within 7 days.

  20. Participation in another investigational protocol 21. Unwillingness or inability to comply with any protocol requirements 22. Pregnant or nursing 23. Extensive prior dissection from a coronary guidewire use 24. Drug abuse or alcoholism. 25. Patients under custodial care. 26. Bleeding diathesis or coagulation disorder; 27. Kawasaki's disease or other vasculitis.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
lack of device related major adverse event | 30 days
  . 30-day Lack of device-related Major Adverse Cardiac Event Rate (MACE) at the site of target coronary lesion and/or its proximal reference segment.
  Time Frame:

SECONDARY OUTCOMES:
Maneuverability of the NovaCross ™ up to the occlusion and safe withdrawal | During Procedure
  Maneuverability of the NovaCross ™ up to the occlusion and safe withdrawal.The ability to cross the lesion with a guidewire in the true lumen, effectively dilate the CTO lesion and place a coronary stent with residual lumen stenosis of less than 30% and restoring antegrade TIMI 3 flow.

CONTACTS AND LOCATIONS:
Overall Officials: Chaim - Lotan, MD, Principal Investigator — Hadassah Ein Karem, Jerusalem Israel
Locations (1):
- Hadasa Ei Karem, Jerusalem, Israel, Israel